CLINICAL TRIAL: NCT06438731
Title: The Effect of Breast Milk and Knitted Octopus on the Pain Caused by Orogastric Tube Insertion in Preterm Newborns
Brief Title: Comparison of Two Methods in Pain Caused by Orogastric Tube Placement in Preterm Newborns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Melek Nur Guzel, researcher, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AIBU-SBF-MG-01
Record Dates: First submitted 2024-05-27; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: Pain; Knitted Octopus; Orogastric Tube; Breast Milk; Preterm
MeSH Terms: conditions — Pain; Premature Birth | interventions — Milk, Human

STUDY DESIGN:
Intervention Model Description: Breast Mılk, Knıtted Octopus And Control Group
Who Masked: Participant
Masking Description: Single blinding (participants) will be used in the study. Participants will not be informed about which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast Milk Group (Active Comparator): Preterm newborns in this group will be administered their own mother's milk with a sterile syringe as 1 ml single dose 2 minutes before orogastric tube insertion. During administration, the baby will not be allowed to suck the tip of the syringe and breast milk will be dripped onto the tongue. Nothing oral will be given 30 minutes before the procedure.
  Interventions: Other: BREAST MILK
- Knitted Octopus Group (Active Comparator): The knitted octopus method will be applied to preterm newborns in this group before orogastric tube insertion. The arms of the knitted octopus will wrap around the baby's arms and legs, and its head will be on the baby's body.
  Interventions: Other: KNITTED OCTOPUS
- Control Group (No Intervention): For preterm newborns in this group, no method will be applied before orogastric tube insertion and routine procedures will be performed.

INTERVENTIONS:
Other: BREAST MILK — The preterm will be monitored for 5 minutes before birth, during the procedure cycle, and then by camera recording for 5 minutes
  Arms: Breast Milk Group
Other: KNITTED OCTOPUS — The preterm will be monitored for 5 minutes before birth, during the procedure cycle, and then by camera recording for 5 minutes
  Arms: Knitted Octopus Group

SUMMARY:
Aim : This study will be conducted to determine the effect of breast milk and knitted octopus in reducing pain caused by routine orogastric tube insertion in preterm newborns.

Method : This study was planned as a randomized controlled trial. The study group will consist of 66 preterms with a gestational age of 32-34 weeks fed by orogastric tube. Informed Consent Form, Preterm Newborn Introduction Form, Physiologic Parameters Measurement Form and Premature Infant Pain Profile (PIPP) will be used in the study. The research will be conducted in the Neonatal Intensive Care Unit of a university hospital in Denizli province. Newborns in the breast milk group will be given oral breast milk before the procedure. Newborns in the knitted octopus group will be provided with the octopus touching various parts of their bodies as a tactile stimulation before the procedure. No intervention will be performed on newborns in the control group. Data will be obtained by the researcher from camera recording and patient file. In evaluating the data, continuous variables will be given as mean ± standard deviation and categorical variables will be given as number and percentage. Parametric and non-parametric tests will be used to examine the differences between groups.

Hypothesis: It is expected to contribute to the development of a new approach in the pain management of preterm newborns by evaluating the effectiveness of breast milk and knitted octopus in reducing the pain caused by orogastric tube insertion in preterm newborns.

DETAILED DESCRIPTION:
İNTRODUCTİON Preterm babies experience many problems in the postnatal period because they are anatomically and physiologically immature.Nutritional problems have an important place among these problems.In the first days of life, they are fed enterally via orogastric tube. Enteral nutrition is the process of giving the newborn's nutrition through a nasogastric (NG), orogastric (OG) or transpyloric tube.Baby feeding tube insertion causes pain.Although in the past years it was said that the newborn did not feel pain, the prenatal starts to feel it from the 20th week. When pain is not detected, the growth and development of the newborn is negatively affected.There are pharmacological and non-pharmacological methods in pain management.

Touch is considered the most basic communication and is well developed. Breast milk increases immunity and ensures growth and development.The sense of taste is highly developed even in premature babies.

There is no study in the literature comparing breast milk and the knitting octopus method together.Considering that orogastric tube application in newborns is a common clinical practice, it is important to minimize the side effects of this treatment method and increase the comfort of babies.

Aim of the study: This study will be conducted to determine the effect of breast milk and knitted octopus in reducing pain caused by routine orogastric tube insertion in preterm neonates.

Materials and Methods

Type of Research The research will be conducted as a randomized controlled study.

Location Characteristics and Time Where the Research Was Conducted The study will be conducted between March 2024 and March 2026 in preterm neonates who received an orogastric tube in the neonatal intensive care unit of a university hospital in a province in the western region of Turkey. In the hospital where the study was conducted, there are level 3, level 2 and maternal adaptation room in the neonatal intensive care unit. Approximately 31 nurses and 2 specialist doctors work in the neonatal intensive care unit.

Population and Sample of the Study The study population will consist of newborns who received treatment and care in the Neonatal Intensive Care Unit of a university hospital in a province in the western region of Turkey between March 2024 and March 2026 and who meet the case selection criteria.

The study sample will consist of preterm newborns with a gestational age of 32-34 weeks treated in the Neonatal Intensive Care Unit of the same hospital. Infants fed with orogastric catheter in the neonatal intensive care unit will be included in the sample. The effect size obtained in the reference study was found to be strong (F=0.695) (Şener Taplak and Erdem 2017). Assuming that a lower effect size (F=0.4) could be obtained, as a result of the power analysis performed for 3 groups, it was calculated that 80% power could be obtained at 95% confidence level when at least 66 infants (at least 22 infants for each group) were included in the study.

Randomization Randomization in the research will be provided by the sealed envelope method. In the case of an infant meeting the sampling criteria, after obtaining signed informed consent from the parent, the researcher will give the newborn a letter placed in a sealed envelope and the newborns will be randomly assigned to groups. Which letter will represent which group will be determined at the beginning of the study using the closed opaque envelope method. Accordingly, letter C will be used for the control group, letter B for the knitted octopus group and letter A for the breast milk group.

Blinding Single blinding (participants) will be used in the study. Participants will not be informed about which group they are in.

Research Inclusion Criteria

* Gestational week between 32-34 weeks
* Postnatal age ≤ 37 weeks
* Having breast milk
* Weighing 1000 grams or more
* Spontaneous breathing
* Being fed with an orogastric tube
* Not being exposed to a painful procedure at least half an hour before the interventions
* Parental consent for the newborn to participate in the study

Criteria for Exclusion from the Study

* Having received ventilator support (may have received it before)
* Any congenital anomaly of the face or oral cavity
* Grade 3 and 4 intraventricular hemorrhage
* Taking opioid or non-opioid analgesics
* Repeated orogastric tube placement

Application

After the parents accept the study and complete the Informed Consent Form, the Preterm Newborn Introduction Form will be completed.Pain level will be evaluated by interpreting the camera image in accordance with the physiologic parameters measurement form and Premature Infant Pain Profile.

Orogastric tube application is applied in neonatal intensive care unit to babies who cannot take by mouth.Orogastric tubes can be changed daily or during the day according to the needs of the newborn.

Since the pain level of breast milk, knitted octopus and control group will be recorded with a camera during the orogastric catheter insertion procedure, the procedure will be performed only once.

Breast Milk Group Preterm newborns in this group will be administered their own mother's milk with a sterile syringe as 1 ml single dose 2 minutes before orogastric tube insertion. During administration, the baby will not be allowed to suck the tip of the syringe and breast milk will be dripped onto the tongue. Nothing oral will be given 30 minutes before the procedure. Preterm newborn will be monitored by camera recording for 5 minutes before, during and 5 minutes after the procedure.

Knitted Octopus Group The knitted octopus method will be applied to preterm newborns in this group before orogastric tube insertion. The arms of the knitted octopus will wrap around the baby's arms and legs, and its head will be on the baby's body. The preterm newborn will be monitored by camera recording for 5 minutes before the procedure, and for 5 minutes during and after the procedure.

Control Group For preterm newborns in this group, no method will be applied before orogastric tube insertion and routine procedures will be performed. The preterm will be monitored for 5 minutes before birth, during the procedure cycle, and then by camera recording for 5 minutes.

Data Collection Tools

Informed Consent Form (Annex 1) It will include information such as the purpose of the research, that participation is voluntary, and that personal information will be kept confidential.

Preterm Newborn Introduction Form (Annex 2) The form prepared by the researcher will include the group in which the newborn is included, mode of delivery, 1st and 5th minute apgar score, birth weight, gender, gestational age, postnatal age and duration of orogastric catheter insertion.

Physiological Parameters Measurement Form (Annex 3) This form prepared by the researcher will help evaluate the pain, heart rate and oxygen saturation value while the orogastric tube is inserted. This form is preterm It was created to record the baby's heart rate and oxygen saturation value. During orogastric tube insertion, heart rate and oxygen saturation will be recorded 1 minute before the procedure, during the procedure, and 1 and 2 minutes after the procedure

Premature Infant Pain Profile (PIPP) (Appendix 4) Stevens et al. Premature Baby Pain Scale ( Premature ) by (1996) baby Pain Profile - PIPP) has been developed. Stevens et al. (1996) found the Cronbach alpha value to be 0.71 for all items of the PIPP. (Apaydın Cırık 2019). Turkish validity and reliability study was conducted by Akcan and Yiğit (2015). In the study conducted by Akcan and Yiğit on preterm newborns between 26-36 weeks and 0-28 days old, the PIPP score was 4.0, 15.0 and 7.0 before, during and after invasive intervention. They found consistency between PIPP elements to be between 0.68 and 0.78, and homogeneity to be between 0.48 and 0.95 (Akcan and Yiğit 2015).

In order to evaluate the baby's pain, the PIPP scale questions 7 items such as gestational age, behavioral status, highest heart rate value, lowest oxygen saturation value, forehead wrinkling, squinting of the eyes and widening of the nose wings. Each item; It is scored as 0, 1, 2 and 3, from best to worst. According to the Premature Baby Pain Profile, the baby's pain is evaluated based on the total score. Accordingly, the highest is 21 points and the lowest is 0 points. If the Premature Baby Pain Profile is between 0 and 6 points, the pain is considered mild, between 7 and 12 points, it is considered moderate, and between 13 and 21 points, the pain is considered severe.

Preterm recorded with a camera device The behavioral responses of newborns at the 1st minute before the procedure , during the procedure, and at the 1st and 2nd minute after the procedure will be evaluated with PIPP.

Tools and equipment to be used in the study; Camera Pulse Oximeter Device Oxygen Saturation Probe Injector Knitted Octopus

Knitted octopus: The material must be washable and sterilizable so that the octopus can share the same space with the babies in the incubator, octopus parts such as eyes and mouth should be sewn, not plastic. Knitted octopuses must be crocheted from cotton yarns (100% cotton), 8/4 or 8/8 cotton, acrylic (washable at 60°C and must be hypoallergenic), fiber-filled 3.0 mm or 3.5 mm in size and protected from accidents . To avoid this, it is recommended that the tentacles (Junior &Coelho 2020) be 20 to 22 centimeters long and consist of 8 tentacles with a head of 8 to 10 centimeters (Siqueira 2019). In line with this data, it is planned to knit 3 octopuses initially and use them alternately after appropriate cleaning methods.

Ethical Dimension Ethical approval for the conduct of the research was received from Pamukkale University Non-Interventional Clinical Research Ethics Committee (10.01.2024 Decision number: E-60116787-020-474228) ; Institutional permission was obtained from Pamukkale University Hospital for the intensive care unit where the study will be conducted.

Analysis Data will be analyzed with the SPSS 25.0 (IBM SPSS Statistics 25 software (Armonk, NY: IBM Corp.)) package program.Continuous variables will be given as mean ± standard deviation and categorical variables will be given as number and percentage. In examining the differences between groups, the significance test of the difference between two means and one-way analysis of variance will be used when parametric test assumptions are met, and Mann Whitney U test and Kruskal Wallis Analysis of Variance will be used when parametric test assumptions are not met. Differences between categorical variables will be examined with Chi square analysis. p <0.05 will be considered statistically significant.

Hypothesis:

This study aims to investigate the effect of breast milk and knitted octopus on pain caused by orogastric tube insertion in premature newborns.

However, there is no study in the literature comparing breast milk and the octopus knitting method together. Considering that orogastric tube application in newborns is a common clinical practice, it is important to minimize the side effects of this treatment method and increase the comfort of babies. After the completion of the study, it is thought that breast milk and knitted octopus will reduce the pain during orogastric tube insertion and can be used as a common practice in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Gestational week between 32-34 weeks
* Postnatal age ≤ 37 weeks
* Having breast milk
* Weighing 1000 grams or more
* Spontaneous breathing
* Being fed with an orogastric tube
* Not being exposed to a painful procedure at least half an hour before the interventions
* Parental consent for the newborn to participate in the study

Exclusion Criteria:

* Having received ventilator support (may have received it before)
* Any congenital anomaly of the face or oral cavity
* Grade 3 and 4 intraventricular hemorrhage
* Taking opioid or non-opioid analgesics
* Repeated orogastric tube placement

Ages: 32 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Premature Infant Pain Profile (PIPP) | one year
  In order to evaluate the baby's pain, the PIPP scale questions 7 items such as gestational age, behavioral status, highest heart rate value, lowest oxygen saturation value, forehead wrinkling, squinting of the eyes and widening of the nose wings. Each item; It is scored as 0, 1, 2 and 3, from best to worst. According to the Premature Baby Pain Profile, the baby's pain is evaluated based on the total score. Accordingly, the highest is 21 points and the lowest is 0 points. If the Premature Baby Pain Profile is between 0 and 6 points, the pain is considered mild, between 7 and 12 points, it is considered moderate, and between 13 and 21 points, the pain is considered severe.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Nur GÜZEL, Principal Investigator — BAĞLANTISIZ; Sebahat ALTUNDAĞ, Study Director — BAĞLANTISIZ
Locations (1):
- Pamukkale University Hospital, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akkaya-Gul A, Ozyazicioglu N. Effect of pacifier and pacifier with dextrose in reducing pain during orogastric tube insertion in newborns: a randomized controlled trial. J Perinatol. 2024 May;44(5):717-723. doi: 10.1038/s41372-024-01948-w. Epub 2024 Mar 29. PMID 38553602
- [Background] Sener Taplak A, Erdem E. A Comparison of Breast Milk and Sucrose in Reducing Neonatal Pain During Eye Exam for Retinopathy of Prematurity. Breastfeed Med. 2017 Jun;12:305-310. doi: 10.1089/bfm.2016.0122. Epub 2017 Apr 17. PMID 28414522
- [Background] Srivastava G, Garg A, Chhavi N, Faridi M. Effect of kangaroo mother care on pain during orogastric tube insertion in low-birthweight newborns: An open label, randomised trial. J Paediatr Child Health. 2022 Dec;58(12):2248-2253. doi: 10.1111/jpc.16212. Epub 2022 Sep 21. PMID 36131630
- [Background] Bueno M. Combined non-pharmacological interventions minimise pain during orogastric tube insertion in preterm neonates. Evid Based Nurs. 2020 Aug 12:ebnurs-2020-103267. doi: 10.1136/ebnurs-2020-103267. Online ahead of print. No abstract available. PMID 32796001
- [Background] Calik C, Esenay F. The clinical effect of pacifier use on orogastric tube-fed preterm infants: A randomized controlled trial. J Pak Med Assoc. 2019 Jun;69(6):771-776. PMID 31189280
- See also: THE EFFECT OF BREAST MILKING, WRAPPING AND FETAL POSITIONING METHODS IN REDUCING THE PAIN DUE TO OROGASTRIC TUBE INSERTION IN PRETERM NEWBORN. — http://acikerisim.akdeniz.edu.tr/bitstream/handle/123456789/4204/T05378.pdf?sequence=1&isAllowed=y
- See also: Effect of Mothers' Heartbeats Combined with Swaddling Technique on Orogastric Tube Insertion Pain among Preterm Neonates — https://ejhc.journals.ekb.eg/article_228203_86b0d67cb5eba3c36c41dfacc2c9dca4.pdf
- See also: Crochet octopuses help soothe premature babies in Araçatuba — https://g1.globo.com/sao-paulo/sao-jose-do-rio-preto-aracatuba/noticia/polvos-de-croche-ajudam-a-acalmar-bebes-prematuros-em-aracatuba.ghtml
- See also: Use of crochet octopus for premature babies in the neonatal unit: an electronic news analysis — https://www.e-publicacoes.uerj.br/index.php/enfermagemuerj/article/download/43566/33044